CLINICAL TRIAL: NCT02482233
Title: A Pilot Randomized Controlled Clinical Trial - "Electronic Nicotine Delivery Device (E-cigarette) for Perioperative Smoking Cessation in Veterans"
Brief Title: The END Perioperative Smoking Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-15274
Record Dates: First submitted 2015-06-17; First posted 2015-06-26 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Smoking; Nicotine Addiction; Surgery
Keywords: electronic cigarette; nicotine replacement therapy; smoking cessation; perioperative
MeSH Terms: conditions — Smoking; Tobacco Use Disorder; Vaping; Smoking Cessation | interventions — Nicotine Replacement Therapy; Nicotine; Tobacco Use Cessation Devices; Crisis Intervention

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ENDD (Experimental): 6-week supply of disposable "NJOY" ENDDs (e-cigarettes)
  * the number of e-cigarettes will be determined by equating the number of e-cigarettes to the number of cigarettes smoked per day (1 pack per day = 2 e-cigarettes per day = 14 e-cigarettes/week)
  * veterans will be given detailed instructions for use and also instructed to start with the high nicotine content (4.5%) strength for three weeks, then decrease to the low nicotine content (2.4%) for two weeks, then switch to nicotine-free for the final week
  Both groups will receive:
  i) referral to the California Smokers' Helpline, ii) brief advice lasting less than 2 minutes, iii) a brochure from the ASA about quitting smoking before surgery
  Interventions: Behavioral: ENDD (NJOY); Behavioral: telephone counseling; Behavioral: brief advice; Behavioral: brochure
- NRT (NicoDerm CQ) (Active Comparator): A prescription for 6 weeks of transdermal nicotine replacement (on-formulary at the VA) in the following doses: For smokers of 10 cigarettes per day or more, a 3-week supply of 21 mg/d, 1-week supply of 14 mg/d, 1-week supply of 7 mg/d, and 1-week of 0mg/d. Smokers of <10 cigarettes per day, 3 weeks of 14 mg/d patches 2 weeks of 7 mg/d patches, and 1-week of 0mg/d.
  Both groups will receive:
  i) referral to the California Smokers' Helpline, ii) brief advice lasting less than 2 minutes, iii) a brochure from the ASA about quitting smoking before surgery
  Interventions: Drug: NRT (NicoDerm CQ); Behavioral: telephone counseling; Behavioral: brief advice; Behavioral: brochure

INTERVENTIONS:
Behavioral: ENDD (NJOY) — As described above.
  Other Names: electronic nicotine delivery device; NJOY e-cigarettes
  Arms: ENDD
Drug: NRT (NicoDerm CQ) — As described above.
  Other Names: nicotine patch
  Arms: NRT (NicoDerm CQ)
Behavioral: telephone counseling — Referral to the California Smokers' Helpline. California Smokers' Helpline will call the patient 4 times, or as agreed upon by the patient.
Behavioral: brief advice — Brief advice lasting less than 2 minutes will be delivered by the research assistant, investigator, or healthcare provider. The advice will be similar to the following statement (customized as needed to the patient): "The most important advice I can give you is that quitting smoking is the number one thing you can do for your health and to prepare yourself for surgery. Quitting smoking before surgery may improve your chances of healing quickly. There's evidence that the longer you quit before your surgery, the fewer complications you'll have. I encourage you to make use of the resources that have been provided to you to help you quit and set your quit date for as soon as possible."
Behavioral: brochure — A brochure from the ASA (American Society of Anesthesiologists) about quitting smoking before surgery.
  Available free from the ASA: http://ecommerce.asahq.org/publicationsAndServices/PatientBrochure_%20For%20Posting.pdf

SUMMARY:
The purpose of this pilot randomized trial is to determine the feasibility of e-cigarettes and telephone counselling (compared to transdermal nicotine replacement and telephone counselling) as a harm-reduction tool that may lead to increased smoking cessation in the perioperative setting in smokers presenting for elective surgery at the San Francisco Veterans Affairs Medical Center. Secondary outcomes include acceptability of e-cigarettes over transdermal nicotine replacement, length-of-stay in the post-anesthesia care unit, hospital length-of-stay, postoperative complications within the first 30-days, and smoking status 8-weeks after randomization. This pilot study is designed to provide the preliminary data necessary to plan and fund a larger-scale randomized clinical trial that will assess the utility of e-cigarettes in achieving smoking cessation perioperatively. Our ultimate goal is to add to the limited existing data on the safety and efficacy of e-cigarette use in smoking cessation, specifically in the perioperative setting where the risks of continued smoking are great and the motivation to stop is high.

DETAILED DESCRIPTION:
It is well-known that smokers suffer more complications and higher risk of mortality after surgery than non-smokers. Despite this knowledge, it is unclear what clinicians can do to minimize this risk. Surgery represents a 'teachable moment' that might encourage smokers to engage in permanent cessation. Several small trials have shown that smoking cessation interventions can increase smoking cessation and reduce postoperative complications, particularly wound-healing complications, which can have an absolute risk reduction of up to 25%. Smoking cessation initiated in the perioperative period can also promote long-term smoking cessation. Despite the benefits of comprehensive smoking cessation interventions including nicotine replacement therapy, current standard of care at the SFVAMC does not routinely include specific preoperative smoking cessation pharmacotherapy or counselling. Although there is an urgent need for more data, e-cigarettes have been proposed as an alternative to nicotine replacement therapy that are at least as effective for smoking cessation, and may be more acceptable to some patients.

The main hypothesis of this pilot study is that the use of e-cigarettes and telephone counselling, compared to telephone counselling and transdermal nicotine replacement, in the perioperative period results in increased smoking cessation on the day of surgery and at 8-weeks after randomization in smokers presenting for elective surgery. As secondary hypotheses, the study will also assess the acceptability of e-cigarettes versus nicotine patches, postoperative complications within the first 30-days, length-of-stay in the PACU and hospital length-of-stay. The investigators will examine the above hypotheses through the following aims:

" Aim 1) To determine how e-cigarettes plus counselling compare to transdermal nicotine replacement plus counselling for the achievement of smoking cessation, when introduced prior to elective surgery in veterans.

The investigators plan to carry-out a pilot randomized controlled trial with parallel design comparing e-cigarettes and telephone counselling with transdermal nicotine replacement and telephone counselling. Our primary outcome is smoking cessation on the day of surgery, as confirmed biochemically by exhaled carbon monoxide. Smoking reduction (self-reported cigarettes per day) of 50% or more and bedside spirometry readings will be assessed as secondary outcomes.

" Aim 2) To determine the acceptability of e-cigarettes amongst veterans as an aid for smoking cessation and to determine the feasibility of recruitment, randomization, and follow-up procedures in preparation for large-scale trial.

Through implementation of this pilot trial, the investigators will determine the feasibility and acceptability of e-cigarettes for smoking cessation perioperatively in the veteran population and obtain the preliminary data necessary to run a larger trial on the effectiveness of e-cigarettes as a perioperative smoking cessation aid.

" Aim 3) To determine the safety of e-cigarettes as a harm reduction strategy to achieve short-term perioperative smoking cessation.

The investigators plan to improve the overall knowledge of the safety of short-term e-cigarettes use through careful surveillance for adverse events and side effects.

" Aim 4) To determine if e-cigarette use preoperatively is associated with a lower risk of complications postoperatively.

The investigators plan to measure the following secondary outcomes: postoperative complications and mortality within the first 30 days, post-anesthesia care unit (PACU) length-of-stay, and hospital length-of-stay. This will help us understand if e-cigarettes have the potential to be used for harm-reduction perioperatively.

ELIGIBILITY:
Inclusion Criteria:

* adults (age >18)
* any gender
* scheduled to undergo elective surgery at the San Francisco Veterans Affairs Medical Center (SFVAMC)
* daily smoker, based on self-report of at least 2 cigarettes/day and having smoked in the last 7 days
* presenting to the anesthesia preoperative (APO) clinic at least 3 days preoperatively

Exclusion Criteria:

* emergency surgery (booked <24 hours preoperatively)
* consumers of non-cigarette forms of tobacco only (pipe, smokeless tobacco) or marijuana only
* already enrolled in a smoking cessation trial
* current smoking cessation pharmacotherapy
* daily user of e-cigarettes
* previous adverse reaction to e-cigarette or transdermal nicotine
* poor proficiency of English language¸as indicated by need for an interpreter (including family members) at the preadmission visit
* lacking capacity for consent (e.g. due to mental illness or dementia), as indicated by consent for surgery and other medical procedures being obtained from a substitute decision maker
* pregnant or breastfeeding
* unstable cardiac condition (unstable angina, unstable arrhythmia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Lee, MD, MAS, Principal Investigator — UCSF / SFVAMC
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

REFERENCES:
- [Result] Lee SM, Tenney R, Wallace AW, Arjomandi M. E-cigarettes versus nicotine patches for perioperative smoking cessation: a pilot randomized trial. PeerJ. 2018 Sep 28;6:e5609. doi: 10.7717/peerj.5609. eCollection 2018. PMID 30280019
- See also: Full peer-reviewed results — https://peerj.com/articles/5609/

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine Replacement Patch Group (Control): Patients randomized to the NRT group received a 6-week supply of NicodermCQ patches (5 weeks) and placebo patches (1 week) appropriate to baseline nicotine consumption.
- Electronic Cigarette (END) Group: Those allocated to the END group received a 6-week supply of NJOY e-cigarettes (Scottsdale, AZ, USA) and were instructed to use the Bold (4.5%) e-cigarettes ad libitum for 3 weeks, the Gold (2.4%) e-cigarettes ad libitum for 2 weeks and the Study (0%) ecigarettes ad libitum for the final week.
Period: Overall Study
Arm/Group | Nicotine Replacement Patch Group (Control) | Electronic Cigarette (END) Group
Started | 10 | 20
Completed | 9 | 19
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Nicotine Replacement Therapy (NRT); Electronic Cigarette (END): As described above
- Total: Total of all reporting groups
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END) | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (10.6) | 54 (12.7) | 54 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 9 | 18 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 10 | 18 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 5 | 11 | 16
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 3 | 3
Day seen prior to surgery [Mean (Standard Deviation); unit: days] | 16.5 (9.5) | 11.2 (7.9) | 13.0 (8.4)
Diabetes [Count of Participants; unit: Participants] | 0 | 2 | 2
Hypertension [Count of Participants; unit: Participants] | 3 | 7 | 10
Heart disease [Count of Participants; unit: Participants] | 0 | 1 | 1
COPD [Count of Participants; unit: Participants] | 1 | 6 | 7
Cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes] | 10.8 (6.6) | 15.3 (10.5) | 13.8 (9.2)
Number of years smoking [Mean (Standard Deviation); unit: years] | 32 (16.4) | 32 (15.6) | 32 (15.9)
Fagerstrom score [Mean (Standard Deviation); unit: units on a scale out of 10 min 1 max 10] — Fagerstrom is a validated scale for nicotine dependence. Higher score indicates more dependence. (min 1 max 10) 1-2 = low, 3-4 = low/mod, 5-7 = moderate, 8+ = high dependence
  units on a scale out of 10 min 1 max 10 | 2.5 (0.9) | 3.7 (2.6) | 3.3 (2.0)
Salivary cotinine (ng/ml) [Mean (Standard Deviation); unit: ng/ml] | 130.1 (75.3) | 209.6 (110.3) | 183.1 (98.6)
Exhaled CO (ppm) [Mean (Standard Deviation); unit: ppm] | 16.1 (7.7) | 21.7 (11.5) | 19.8 (10.2)
FEV1 (L) [Mean (Standard Deviation); unit: L] | 3.14 (1.35) | 2.78 (1.11) | 2.9 (1.2)
FVC (L) [Mean (Standard Deviation); unit: L] | 3.52 (1.28) | 4.03 (1.32) | 3.9 (1.31)
FEV1/FVC (%) [Mean (Standard Deviation); unit: percent] | 105 (81.3) | 68.2 (13.0) | 80.5 (35.8)

OUTCOME MEASURES:

1. Primary Outcome: Smoking Status on the Day of Surgery (48-hour Point-prevalence Abstinence), by Self-report and Confirmed With Exhaled Carbon Monoxide (CO)
Description: Confirmed abstinent. Abstinence confirmed with exhaled carbon monoxoide <10ppm.
  Time Frame depends on date of preadmission clinic visit
Time Frame: day of surgery (expected average around 1-2 weeks after enrollment/randomization)
Measure: Count of Participants; unit: Participants
Groups:
- Nicotine Replacement Therapy (NRT); Electronic Cigarette (END): As above
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 10 | 20
Participants | 2 | 3

2. Secondary Outcome: Frequency of Use of Product - Number Reporting Use Daily or Most Days
Description: how often product (e-cigarette or patch) was used (everyday except while hospitalized, most days, a few times a week, once a week, less than once a week, not at all)
  Result reported is those that used the product daily or most days
Time Frame: 8-weeks
Population: in-person visit at 8-weeks, or make-up phone call if unavailable in-person
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 10 | 19
Participants | 6 | 16

3. Secondary Outcome: Report of How Helpful the Product Was for Quitting
Description: 7-point likert scale (strongly disagree to strongly agree)
  1. strongly disagree
  2. disagree
  3. disagree somewhat
  4. neither agree nor disagree
  5. agree somewhat
  6. agree
  7. strongly agree
Time Frame: 8-weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale out of 7
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 10 | 19
units on a scale out of 7 | 5 [3 to 7] | 6 [4 to 7]

4. Secondary Outcome: How Satisfied the Patient Was With the Product (E-cigarette or Patch)
Description: as for outcome 3
Time Frame: 8-weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale out of 7
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 10 | 19
units on a scale out of 7 | 5 [3 to 6] | 5.5 [2.5 to 7]

5. Secondary Outcome: How Likely the Patient Would be to Recommend the Product (E-cigarette or Patch) to Others
Description: as for outcome 3
Time Frame: 8-weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale out of 7
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 10 | 19
units on a scale out of 7 | 7 [6 to 7] | 6 [5 to 7]

6. Secondary Outcome: Smoking Status 8-weeks After Randomization (Confirmed by Exhaled CO)
Description: by self-report and confirmed by exhaled CO<10ppm - confirmed abstinent
Time Frame: 8-weeks
Population: Those lost to follow-up assumed to still be smoking (1 in NRT group). Those who had telephone interview were unable to have exhaled CO verification (n=1 in NRT group, n=2 in END group). Since they were not verified by exhaled CO, they were not considered abstinent.
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 9 | 20
Participants | 0 | 3

7. Secondary Outcome: Smoking Reduction
Description: 50% or less regular cigarette use compared to baseline as determined by asking participants to self-report daily cigarette use in cigarettes per day at each time point.
Time Frame: on day of surgery and 8-weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 10 | 20
Participants | 7 | 13

8. Secondary Outcome: Number of Participants With Dual Use
Description: use of both regular and e-cigarettes concurrently
Time Frame: on day of surgery and 8-weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 10 | 20
Participants | 3 | 2

9. Secondary Outcome: Spirometry - FEV1/FVC Change
Description: Change in FEV1/FVC from baseline to day of surgery / 8-weeks. FEV1/FVC is expressed in percent. For example, if FEV1/FVC was 75%, 80%, and 85% at baseline, day of surgery and 8-weeks, result is reported as change in FEV1/FVC being +5% and +10% for day of surgery and 8-weeks respectively.
Time Frame: day of surgery and 8-weeks
Measure: Mean (Standard Deviation); unit: percent (change from baseline)
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 10 | 18
percent (change from baseline)
  FEV1/FVC on day of surgery compared to baseline | -32.2 (74) | -1.6 (8.2)
  FEV1/FVC at 8 weeks compared to baseline | -38.1 (79.2) | 2.0 (10.5)

10. Secondary Outcome: Spirometry - FEV1
Description: change in FEV1 (mL) compared to baseline
Time Frame: day of surgery and 8-weeks
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 10 | 18
mL
  change in FEV1 day of surgery | -236 (585) | -163 (549)
  change in FEV1 8-weeks | -300 (497) | 292 (503)

11. Secondary Outcome: Cotinine Level (Change in)
Description: salivary
Time Frame: day of surgery and 8-weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 10 | 18
ng/ml
  day of surgery | 106 (137) | 19 (119)
  8-weeks | 34 (89) | -48 (103)

12. Secondary Outcome: Number of Participants With Postoperative Complications (Composite)
Description: by chart review - research assistant or investigator examined notes and investigations postoperatively for complications by telephone self-report - patients were asked open-ended question about whether they experienced any postoperative complications
Time Frame: 30-days postop
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 10 | 19
Participants
  by chart review | 6 | 5
  by telephone self-report | 2 | 5

13. Secondary Outcome: Long-term Smoking Status - Use of Conventional Cigarettes
Description: by self-report (7-day point prevalence)
Time Frame: 6 months
Population: those lost assumed to still be smoking
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 9 | 20
Participants | 1 | 5

14. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: all patients will be asked about adverse events each time they are contacted (day of surgery, 30-days postoperatively, and 8-weeks after randomization), and they will also be able to call to report adverse events to the study team any time during the study.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 9 | 19
Participants
  any adverse event | 3 | 10
  moderate adverse event (required intervention) | 1 | 1

15. Secondary Outcome: Number of Participants Postoperative Complications (Composite)
Description: by telephone self-report
Time Frame: 30-days postop
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
Number analyzed (Participants) | 10 | 19
Participants | 2 | 5

ADVERSE EVENTS:
Arm/Group | Nicotine Replacement Therapy (NRT) | Electronic Cigarette (END)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 6/10 | 10/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Replacement Therapy (NRT) (N=10) | Electronic Cigarette (END) (N=20)
Headache (Nervous system disorders) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5)
Dry cough (persistent) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dry cough (intermittent) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
palpitations (Cardiac disorders) | 2 (2) | 0 (0)
throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
skin irritation (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
other (General disorders) | 6 (6) | 7 (7) — includes (for NRT group) irritable mood, patch not sticking properly, increased cravings, jitteriness, diarrhea, dry mouth, anxiety, sleepiness and (for END group) wheezing, productive cough, choking sense, poor appetite, burning sensation, lip burn

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes